CLINICAL TRIAL: NCT06768606
Title: Single Arm Study of a Novel Social-emotional Learning Curriculum in STEM-based After-school Program for Youth
Brief Title: Feasibility of a Social-emotional Learning Curriculum in a STEM-based After-school Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Brendan Andrade, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024/159
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Feasibility Study; Social-emotional Learning Curriculum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: Social-emotional learning curriculum (Experimental): This is the only group delivering the EMPOWER social-emotional learning curriculum.
  Interventions: Behavioral: EMPOWER Social-emotional learning curriculum

INTERVENTIONS:
Behavioral: EMPOWER Social-emotional learning curriculum — EMPOWER is a 16-week social-emotional learning curriculum that is integrated into the after-school program context. The STEM Academy program will implement a shortened version of the social-emotional learning curriculum to meet their timelines.

SUMMARY:
The goal of this single arm study is to:

1. primary purpose: to determine the feasibility of a novel social-emotional learning curriculum when implemented in the STEM Academy program at the Visions of Science after school program; 2a. secondary purpose: to determine whether the novel social-emotional learning curriculum has positive effects youth social emotional learning skills; 2b. secondary purpose: to determine whether the novel social-emotional learning curriculum has positive effects on youth resilience and overall functioning.

Participants:

1. Facilitators working with the STEM Academy program at the Visions of Science after school program
2. Youth aged 11-14 who participate in the STEM Academy program at the Visions of Science after school program
3. Parents of youth who participate in the STEM Academy Visions of Science after school program

The main questions this study aims to answer are:

Primary Objectives:

1. Is the novel social-emotional curriculum feasible within the STEM Academy program at the Visions of Science after school program?
2. Is the novel social-emotional curriculum acceptable within the STEM Academy program at the Visions of Science after school program?
3. Is the novel social-emotional curriculum appropriate within the STEM Academy program at the Visions of Science after school program?

Secondary Objectives: Social-emotional learning skills

1. Have youth social-emotional learning skills improved as a result of participating in the novel social-emotional learning curriculum?

Secondary Objectives: Resilience and overall functioning

1. Have youth resilience abilities and overall functioning improved as a result of participating in the novel social-emotional learning program?

Comparator: None

Measures:

Primary Objective: Feasibility

After school program staff participants will be asked to complete:

* 3 feasibility measures (feasibility, acceptability, appropriateness of intervention) after each social-emotional module they complete teaching.
* weekly fidelity checklists to assess feasibility.

Youth participants will be asked to complete:

- the intervention appropriateness measure during the post-curriculum data collection time point.

Secondary Objective: Social-emotional learning skills

After school program staff participants will be asked to complete the following measure pre- and post-curriculum implementation:

- social-emotional learning skills measure for each youth aged 11-14 years in their class.

Youth participants will be asked to complete the following measure pre- and post-curriculum implementation:

- social-emotional learning skills measure Parents participants whose youth are in the intervention arm will be asked to participate in an interview.

Secondary objective: Resilience and overall functioning

After school program staff participants will be asked to complete the follow measures pre- and post-curriculum implementation:

- overall functioning measure for each youth aged 11-14 years in their class.

Youth participants will be asked to complete:

- resilience measure

DETAILED DESCRIPTION:
The EMPOWER project is a community-academic partnership between 2 after school programs (beyond 3:30 and Visions of Science) and a mental health teaching hospital (Centre for Addiction and Mental Health). The main objective of this project is to bolster youth mental well-being by developing a novel social-emotional learning curriculum that after school programs can embed into their existing activities.

The curriculum is designed to improve youth's social emotional learning skills through the integration of short social-emotional learning lessons that are embedded into existing programming within an after-school program. The curriculum is based on the Collaborative for Academic, Social and Emotional Learning's five core SEL competencies that include self-awareness, self-management, social awareness, relationship skills and decision-making.

The investigators have designed a pilot study to test the feasibility and efficacy of the EMPOWER social-emotional learning curriculum. Visions of Science hosts a 14-week program from January - April 2025 called STEM Academy, an after-school science-based program for youth in grades 6-8. We designed a single arm study to assess a shortened and modular use of the EMPOWER social-emotional learning curriculum that is tailored to Visions of Science.

ELIGIBILITY:
INCLUSION:

Youth participants must meet the following inclusion criteria:

1. Must be a youth aged 11-14 years attending the STEM Academy program at the Visions of Science after school program
2. Must sign and date the informed consent form
3. Must speak and understand English

Staff participants must meet the following inclusion criteria:

1. Must be a facilitator of the STEM Academy program at the Visions of Science after school program
2. Must sign and date the informed consent form
3. Must speak and understand English

Caregiver/parent participants must meet the following inclusion criteria:

1. Must be a caregiver/parent of a youth aged 11-14 years attending the STEM Academy program at the Visions of Science after school program. Caregivers/parents whose children decide not to participate in data collection are still able to participate in an interview post-SEL curriculum implementation.
2. Must sign and date the informed consent form
3. Must speak and understand English

EXCLUSION; None

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-21 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by 5-point Likert-type scale | 13 weeks
  Description: Staff will complete the Feasibility of Intervention (Weiner et al., 2017) measure after each social-emotional domain (self-awareness, self-management, social awareness and relationship skills, decision-making) is taught. This is a 4-item, 5-point Likert-type scale that measures a composite feasibility of intervention score.
Acceptability of Intervention | 13 weeks
  Staff in the active intervention arm will complete the Acceptability of Intervention Measure (Weiner et al., 2017) measure after each social-emotional domain (self-awareness, self-management, social awareness and relationship skills, decision-making) is taught. This is a 4-item, 5-point Likert-type scale that measures a composite acceptability of intervention score.
Intervention Appropriateness | 13 weeks
  Staff will complete the Intervention Appropriateness (Weiner et al., 2017) measure after each social-emotional domain (self-awareness, self-management, social awareness and relationship skills, decision-making) is taught. This is a 4-item, 5-point Likert-type scale that measures a composite appropriateness of intervention scale. Youth will complete the intervention appropriateness (Weiner et al., 2017) scale post-SEL curriculum implementation.

SECONDARY OUTCOMES:
Overall functioning | 13 weeks
  KIDSCREEN 10 (Child Public Health, 2023) is a 10-item, 5-point Likert-type scale that measures global quality of life. Staff will complete an adapted version of the KIDSCREEN for each youth they work with (avg. 25 youth/site) pre- and post-EMPOWER SEL curriculum intervention. Youth will complete the KIDSCREEN pre- and post-EMPOWER SEL curriculum intervention.
Resilience | 13 weeks
  Connor-Davidson Resilience Scale (CD-RISC-10; 2007) is a 10-item, 5-point Likert-type scale that measures overall resilience. Youth will complete this measure pre- and post-EMPOWER SEL curriculum intervention.
Social-emotional learning skills | 13 weeks
  The Social Skills Improvement System - Social Emotional Learning (SSIS-SEL Brief Scale; (Elliot et al., 2020) is a 20-item, 4-point Likert-type scale that measures self-awareness, self-management, social awareness, relationship skills, and decision making as a composite score of social-emotional competency. Staff will complete the SSIS-SEL Brief Scale for each youth they work with (avg. 25 youth/site) pre- and post-EMPOWER SEL curriculum intervention. Youth will complete the SSIS-SEL Brief Scale pre- and post-EMPOWER SEL curriculum intervention.

IPD SHARING:
Plan to Share IPD: No